CLINICAL TRIAL: NCT05778500
Title: IMPlementazione di algoRitmi di Assistenza Alla diagnOsi in un Software di Refertazione Computerizzato Che Valuta Anche l'Accuratezza Dell'Esame ECOcardiografico
Brief Title: Algorithms to Improve the Accuracy of the Echocardiographic Report
Acronym: IMPROVE ECO
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Medimatic S.R.L., Genova, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09J002
Record Dates: First submitted 2023-02-24; First posted 2023-03-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Echocardiography
Keywords: Transthoracic echocardiography; Transesophageal echocardiography; Report

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: COMPACS — We will modify the current version of the COMPACS software package to implement several guideline-derived algorithms to help the clinician to reduce diagnostic errors and increase the adherence to current guidelines

SUMMARY:
This observational study aims to improve the accuracy of the report of the echocardiographic study, making it more consistent with the current international guidelines and reducing the diagnostic mistakes in patients undergoing clinically -indicated echocardiography. The main questions it aims to answer are:

* can the addition of automated diagnostic algorithms help to improve the overall accuracy of the echocardiographic report?

ELIGIBILITY:
Inclusion Criteria:

* Having undergone a clinically-indicated echocardiographic study

Exclusion Criteria:

* Denial of the consensus to use individual clinical data for research purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who consecutively undergo an echocardiographic examination
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Inconsistencies between quantitative and qualitative parameters in the report | During analysis of echocardiographic data
  Number of inconsistencies between quantitative and qualitative parameters in the report

SECONDARY OUTCOMES:
Inconsistencies between the clinical diagnosis and clinical guidelines | During analysis of echocardiographic data
  Number of inconsistent clinical diagnoses in the report and indications included in current guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy